CLINICAL TRIAL: NCT02614794
Title: Phase 2 Randomized, Double-Blinded, Controlled Study of Tucatinib vs Placebo in Combination With Capecitabine and Trastuzumab in Patients With Pretreated Unresectable Locally Advanced or Metastatic HER2+ Breast Carcinoma
Brief Title: A Study of Tucatinib vs. Placebo in Combination With Capecitabine & Trastuzumab in Patients With Advanced HER2+ Breast Cancer
Acronym: HER2CLIMB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONT-380-206; 2015-002801-12 (EudraCT Number)
Expanded Access: NCT04220203 (Approved for marketing)
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: HER2 Positive Breast Cancer
Keywords: Tucatinib; Capecitabine; Trastuzumab; Xeloda; Herceptin; Breast Cancer; ARRY-380; ONT-380; HER2 Positive Breast Carcinoma; HER2 Positive Locally Advanced Breast Cancer; HER-2 Positive Breast Cancer; HER-2 Positive Breast Carcinoma; HER-2 Positive Locally Advanced Breast Cancer; Recurrent Breast Carcinoma; Stage IV Breast Cancer; Metastatic Breast Cancer; Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Brain Metastases in Breast Cancer; Asymptomatic Brain Metastases in Breast Cancer; Low Symptomatic Brain Metastases in Breast Cancer; Seattle Genetics
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — tucatinib; Capecitabine; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking applied only during the Double-blind phase of the trial. The Unblinded Phase is open-label.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tucatinib in combination with capecitabine & trastuzumab (Experimental): Tucatinib + capecitabine + trastuzumab
  Interventions: Drug: tucatinib; Drug: capecitabine; Drug: trastuzumab
- Placebo in combination with capecitabine & trastuzumab (Active Comparator): Placebo + capecitabine + trastuzumab
  Interventions: Drug: capecitabine; Drug: trastuzumab; Drug: placebo

INTERVENTIONS:
Drug: tucatinib — 300 mg orally twice daily
  Other Names: ONT-380, ARRY-380
  Arms: Tucatinib in combination with capecitabine & trastuzumab
Drug: capecitabine — 1000 mg/m2 orally twice daily on Days 1-14 of each 21-day cycle
  Other Names: Xeloda
Drug: trastuzumab — 8 mg/kg intravenously (IV) on Day 1 of Cycle 1, followed by 6 mg/kg on Day1 of each 21-day cycle. In regions where approved, trastuzumab may be given at 600mg subcutaneously once every 3-weeks at either study initiation or crossing over from previous IV trastuzumab.
  Other Names: Herceptin, Herceptin Hycleta
Drug: placebo — Oral dose twice daily
  Arms: Placebo in combination with capecitabine & trastuzumab

SUMMARY:
This study is being done to see if tucatinib works better than placebo to help patients who have a specific type of breast cancer called HER2 positive breast carcinoma. The breast cancer in this study is either metastatic (spread into other parts of the body) or cannot be removed completely with surgery. All patients in the study will get capecitabine and trastuzumab, two drugs that are often used to treat this cancer.

There are two parts to this study. The first part of the study is already complete. Patients were randomly assigned to get either tucatinib or placebo (a pill with no medicine). Since this part was "blinded," neither patients nor their doctors knew whether a patient got tucatinib or placebo.

The second part of the study is called the Unblinded Phase. In this part of the study, participants and their doctors know which drugs are being given. Participants who used to get or are currently getting placebo may be able to start taking tucatinib instead.

Each treatment cycle lasts 21 days. Patients will swallow tucatinib pills two times every day. They will swallow capecitabine pills two times a day during the first two weeks of each cycle. Patients will get trastuzumab injections from the study site staff on the first day of every cycle.

DETAILED DESCRIPTION:
This is a randomized, international, multi-center study in patients with progressive unresectable locally advanced or metastatic HER2+ breast cancer who have had prior treatment with trastuzumab, pertuzumab and T-DM1. There are two phases to this trial: the Double-blind Phase and the Unblinded Phase. In the Double-blind phase, participants were randomized in a 2:1 ratio to receive tucatinib or placebo in combination with capecitabine and trastuzumab. In the Unblinded Phase, patients on placebo may be offered tucatinib.

Stratification factors include presence or history of treated or untreated brain metastases or brain lesions of equivocal significance (yes/no), Eastern Cooperative Oncology Group (ECOG) Performance Status (0 vs. 1), and region of world (US vs. Canada vs. Rest of World).

Safety assessments will be performed at a minimum of once every three weeks throughout study treatment and 30 days after the last dose of study drugs. Laboratory assessments will be performed locally at sites. Left ventricular ejection fraction will be assessed by MUGA or ECHO at screening and once every 12 weeks thereafter.

For the blinded phase, contrast brain MRI was performed at baseline. Efficacy assessments (CT of chest, abdomen and pelvis at a minimum) utilized RECIST 1.1 and included patients with evaluable tumors defined as measurable target lesions and non-measurable non-target lesions. RECIST assessment was performed at baseline, every 6 weeks for the first 24 weeks, and then every 9 weeks thereafter. Repeat MRI of the brain was required on this same schedule only in those patients with brain metastases identified at baseline. All treatment decisions were made based upon investigator assessment. All patients underwent a repeat MRI of the brain within 30 days of the end of treatment unless previously performed at time of disease progression.

For the unblinded phase, RECIST assessments will be performed per standard clinical practice as determined by investigator with a maximum interval of 12 weeks.

ELIGIBILITY:
Double-blind Phase Inclusion Criteria

* Histologically confirmed HER2+ breast carcinoma, with HER2+ defined by in situ hybridization (ISH), immunohistochemistry (IHC), or fluorescence in situ hybridization (FISH) methodology
* Received previous treatment with trastuzumab, pertuzumab, and T-DM1
* Progression of unresectable locally advanced or metastatic breast cancer after last systemic therapy (as confirmed by investigator), or be intolerant of last systemic therapy
* Have measurable or non-measurable disease assessable by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate hepatic and renal function and hematologic parameters
* Left ventricular ejection fraction (LVEF) ≥ 50%
* CNS Inclusion - Based on screening brain magnetic resonance imaging (MRI), patients must have one of the following:

  1. No evidence of brain metastases
  2. Untreated brain metastases not needing immediate local therapy
  3. Previously treated brain metastases not needing immediate local therapy

     1. Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy
     2. Patients treated with CNS local therapy for newly identified lesions found on contrast brain MRI performed during screening for this study may be eligible to enroll if the following criteria are met:

     i. Time since whole brain radiation therapy (WBRT) is ≥ 21 days prior to first dose of study treatment, time since stereotactic radiosurgery (SRS) is ≥ 7 days prior to first dose of study treatment, or time since surgical resection is ≥ 28 days.

     ii. Other sites of disease assessable by RECIST 1.1 are present
  4. Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions

Double-blind Phase Exclusion Criteria

* Previously been treated with:

  1. lapatinib within 12 months of starting study treatment (except in cases where lapatinib was given for ≤ 21 days and was discontinued for reasons other than disease progression or toxicity)
  2. neratinib, afatinib, or other investigational HER2/epidermal growth factor receptor (EGFR) or HER2 tyrosine kinase inhibitor (TKI) at any time previously
  3. capecitabine (or other fluoropyrimidine) for metastatic disease except in cases where capecitabine was given for < 21 days and was discontinued for reasons other than disease progression or toxicity. Patients who have received capecitabine for adjuvant or neoadjuvant treatment at least 12 months prior to starting study treatment are eligible.
* Clinically significant cardiopulmonary disease
* Carriers of Hepatitis B or Hepatitis C or have other known chronic liver disease
* Positive for human immunodeficiency virus (HIV)
* Unable for any reason to undergo MRI of the brain
* Have used a strong CYP3A4 or CYP2C8 inhibitor within 5 half-lives of the inhibitor, or a strong CYP3A4 or CYP2C8 inducer within 5 days prior to first dose of study treatment
* Have known dihydropyrimidine dehydrogenase deficiency (DPD)
* CNS Exclusion - Based on screening brain MRI, patients must not have any of the following:

  1. Any untreated brain lesions > 2.0 cm in size, unless approved by medical monitor
  2. Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent)
  3. Any brain lesion thought to require immediate local therapy. Patients who undergo local treatment for such lesions identified by screening contrast brain MRI may still be eligible for the study based on criteria described under CNS inclusion criteria
  4. Known or suspected leptomeningeal disease (LMD)
  5. Poorly controlled seizures Unblinded Phase Crossover Inclusion Criteria - Participants who were randomized to the control arm (placebo + trastuzumab + capecitabine) must meet the following criteria to be eligible to crossover to the experimental arm.
* Have measurable or non-measurable disease assessable by RECIST 1.1
* For patients who were randomized to the control arm and on the long-term follow-up period at the time of crossover screening: have progression of unresectable locally advanced or metastatic breast cancer after last systemic therapy (as confirmed by investigator), or be intolerant of last systemic therapy.
* Have an ECOG Performance Status of 0 or 1
* Have a life expectancy of at least 6 months
* Have adequate hepatic and renal function and hematologic parameters
* Left ventricular ejection fraction (LVEF) ≥ 50%
* CNS Inclusion - Based on screening brain magnetic resonance imaging (MRI), patients must have one of the following:

  i. No evidence of brain metastases ii. Untreated brain metastases not needing immediate local therapy iii. Previously treated brain metastases not needing immediate local therapy
* Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy
* Patients treated with CNS local therapy for newly identified lesions found on contrast brain MRI performed during screening for this study may be eligible to enroll if the following criteria are met:

  1. Time since whole brain radiation therapy (WBRT) is ≥ 21 days prior to first dose of study treatment, time since stereotactic radiosurgery (SRS) is ≥ 7 days prior to first dose of study treatment, or time since surgical resection is ≥ 28 days.
  2. Other sites of disease assessable by RECIST 1.1 are present Unblinded Phase Crossover Exclusion Criteria - Participants who were randomized to the control arm (placebo + trastuzumab + capecitabine) will be excluded from the crossover to the experimental arm for any of the following reasons.
* Discontinuation of study treatment due to an adverse event while on the double-blind phase of the study. If the adverse event leading to discontinuation of study treatment has resolved, the patient may be allowed to crossover with approval from the medical monitor.
* History of exposure to the following cumulative doses of anthracyclines:

  * Doxorubicin > 360 mg/m^2
  * Epirubicin > 720 mg/m^2
  * Mitoxantrone > 120 mg/m^2
  * Idarubicin > 90 mg/m^2
  * Liposomal doxorubicin > 550 mg/m^2
* History of allergic reactions to trastuzumab, capecitabine, or compounds chemically or biologically similar to tucatinib

  o Exceptions for Grade 1 or 2 infusion related reactions to trastuzumab that were successfully managed, or known allergy to one of the excipients in the study drugs
* Have received treatment with any systemic anti-cancer therapy, non-CNS radiation, or experimental agent within 3 weeks prior to start of crossover therapy
* Any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the following exceptions:

  * Alopecia and neuropathy (must have resolved to ≤ Grade 2)
  * CHF (must have been ≤ Grade 1 in severity at the time of occurrence and must have resolved completely)
  * Anemia (must have resolved to ≤ Grade 2)
* Have clinically significant cardiopulmonary disease
* Have known myocardial infarction or unstable angina within 6 months prior to start of crossover therapy
* Require therapy with warfarin or other coumarin derivatives
* Inability to swallow pills or significant gastrointestinal disease which would preclude the adequate oral absorption of medications
* Have used a strong CYP2C8 inhibitor within 5 half-lives of the inhibitor or have used a strong CYP2C8 or CYP34A inducer within 5 days prior to start of the crossover (tucatinib) treatment.
* Known dihydropyrimidine dehydrogenase deficiency
* Unable to undergo contract MRI of the brain
* Have evidence within 2 years prior to start of crossover therapy of another malignancy that required systemic treatment
* CNS Exclusion:
* CNS Exclusion - Based on screening brain MRI, patients must not have any of the following:

  * Any untreated brain lesions > 2.0 cm in size, unless approved by medical monitor
  * Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent)
  * Any brain lesion thought to require immediate local therapy. Patients who undergo local treatment for such lesions identified by screening contrast brain MRI may still be eligible for the study based on criteria described under CNS inclusion criteria
  * Known or suspected leptomeningeal disease (LMD)
  * Poorly controlled seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Ramos, DO, Study Director — Seagen Inc.; Corinna Palanca-Wessels, MD, PhD, Study Director — Seagen Inc.
Locations (176):
- United States (81):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama - Mitchell Cancer Institute, Mobile, Alabama
  - Cancer Treatment Centers of America - Phoenix, Goodyear, Arizona
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - TRIO - Central Regulatory Office, Los Angeles, California
  - UCLA Medical Center / David Geffen School of Medicine, Los Angeles, California
  - Torrance Memorial Physician Network - TRIO, Redondo Beach, California
  - University of California at San Francisco, San Francisco, California
  - Kaiser Permanente San Marcos Medical Offices, San Marcos, California
  - Central Coast Medical Oncology Corporation TRIO, Santa Maria, California
  - Kaiser Permanente Medical Center Northern California, Vallejo, California
  - University of Colorado Hospital / University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Lombardi Cancer Center / Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - South Region, Fort Myers, Florida
  - Memorial Regional Hospital TRIO, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center / Florida, Miami Beach, Florida
  - Orlando Health, Inc. TRIO, Orlando, Florida
  - Florida Cancer Specialists - North Region, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Florida Cancer Specialists - East West Palm Beach, FL (SCRI), West Palm Beach, Florida
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Cancer Treatment Centers of America, Newnan, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Illinois Cancer Specialists / Advocate Lutheran General Hospital, Niles, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Saint Luke's Cancer Institute LLC, Kansas City, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center/ Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Beth Israel, New York, New York
  - New York University (NYU) Cancer Institute, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Services / Brody School of Medicine East Carolina University, Greenville, North Carolina
  - James Cancer Hospital / Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - University of Pennsylvania / Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Cancer Treatment Centers of America / Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Medical University of South Carolina/Hollings Cancer Center, Charleston, South Carolina
  - Wellmont Cancer Institute, Kingsport, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology Methodist, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - The Center for Cancer and Blood Disorders: Fortworth, Fort Worth, Texas
  - Texas Oncology - Houston Memorial City, Houston, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Baylor Clinic, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Paris Regional Medical Center / US Oncology, Paris, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - San Antonio Medical Center Northeast, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - US Oncology Central Regulatory, The Woodlands, Texas
  - Texas Oncology - Deke Slayton Cancer Center, Webster, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Shenandoah Oncology P.C., Winchester, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin
- Australia (9):
  - Austin Hospital, Heidelberg
  - Cabrini Education and Research Precinct, Malvern
  - Peter MacCallum Cancer Centre, Melbourne
  - Breast Cancer Research Centre, Nedlands
  - Mater Hospital, North Sydney
  - Icon Cancer Care South Brisbane, South Brisbane
  - Mater Health Services, South Brisbane
  - Sunshine Hospital, St Albans
  - Westmead Hospital, Westmead
- Austria (4):
  - LKH- Universitat Klinikum Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - KH d. Barmherzigen Schwestern Linz, Linz
  - LKH Salzburg, Universitatsklinikum der PMU, Salzburg
- Belgium (5):
  - AZ Klina, Brasschaat
  - Cliniques Universitaires Saint Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Centre Hospitalier de l'Ardenne, Libramont
  - CHU UCL Namur-Site de Saint Elisabeth, Namur
- Canada (11):
  - Tom Baker Cancer Centre, Calgary
  - University of Alberta / Cross Cancer Institute, Edmonton
  - Queen Elizabeth II Health Sciences Centre, Halifax
  - Jewish General Hospital, Montreal
  - Hopital du Saint-Sacrement, CHU de Quebec-Universite Laval, Québec
  - Allan Blair Cancer Centre, Regina
  - Saskatoon Cancer Centre, Saskatoon
  - H. Bliss Murphy Cancer Centre, St. John's
  - Sunnybrook Health Sciences Centre, Toronto
  - University Health Network, Princess Margaret Hospital, Toronto
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove-oddeleni klinicke hematologie, Hradec Králové
  - Fakultni Nemocnice Olomouc (Fnol) - Onkologicka Klinika, Olomouc
- Denmark (5):
  - Aalborg Universitetshospital, Aalborg
  - Rigs Hospiltalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense C
  - Sygehus Lillebaelt - Vejle Sygehus, Vejle
- France (11):
  - University Hospital of Besancon, Besançon
  - Clinique Victor Hugo, Le Mans
  - Centre Leon Berard - Centre regional de lutte contre le cancer Rhone-Alpes, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institute Curie - Centre de Lutte Contre Le Cancer CLCC de Paris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHU Tours - Hopital Bretonneau, Tours
- Germany (9):
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Koln, Cologne
  - Kliniken Essen-Mitte - Evang. Huyssens-Stiftung, Essen
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) - Onkologisches Zentrum - Interdisziplinaere Klinik und Poliklinik fuer Stammzelltransplantation, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - InVO- Institut fUr Versorgungsforschung in der onkologie GbR, Koblenz
  - HOPE- Onkologisches Zentrum Rotkreuzklinikum, München
  - Sana Klinikum Offenbach GmbH, Offenbach
- Israel (7):
  - Rambam Health Corp., Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (9):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Ospedale di Bolzano, Bolzano
  - Presido Ospedaliero- Senatore Antonio Perrino, Brindisi
  - Ospedale Ramazzini di Carpi, Carpi
  - Ospedale Policlinico San Martino, Genova
  - Istituto Europeo di Oncologia, Milan
  - IRCSS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera S. Maria di Terni, Terni
  - A.O.U. - Ospedali Riuniti di Ancona, Torrette
- Portugal (2):
  - Hospital Cuf Descobertas R. Mario Botas Parque das Nacoes, Lisbon
  - Centro Hospitalar do Porto - Hospital Santo Antonio, Porto
- Spain (10):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Complejo Asistencial Universitario de Leon, León
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Clinico Univ De Santiago De Compostela, Santiago de Compostela
  - Hospital Arnau De Vilanova, Valencia
  - Hospital Clinico Universitario Lozano Blesa de Zaragoza, Zaragoza
- Institute of Oncology of Southern Switzerland, Bellinzona, Switzerland
- United Kingdom (10):
  - Colchester Hospital University NHS Foundation Trust, Colchester
  - The Royal Marsden Hospital, London
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Hospital, UK, Northwood
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Peterborough City Hospital, Peterborough
  - Weston Park Hospital- UK, Sheffield
  - The Royal Marsden Hospital (Surrey), Sutton
  - Royal Cornwall Hospitals NHS Trust, Truro

REFERENCES:
- [Derived] Dai L, Gao T, Guo R, Chen Y, Wang J, Zhou S, Tang Y, Chen D, Huang S. Efficacy and safety of pyrotinib-based regimens in HER2 positive metastatic breast cancer: A retrospective real-world data study. Neoplasia. 2024 Oct;56:101029. doi: 10.1016/j.neo.2024.101029. Epub 2024 Jul 17. PMID 39024777
- [Derived] Lin NU, Murthy RK, Abramson V, Anders C, Bachelot T, Bedard PL, Borges V, Cameron D, Carey LA, Chien AJ, Curigliano G, DiGiovanna MP, Gelmon K, Hortobagyi G, Hurvitz SA, Krop I, Loi S, Loibl S, Mueller V, Oliveira M, Paplomata E, Pegram M, Slamon D, Zelnak A, Ramos J, Feng W, Winer E. Tucatinib vs Placebo, Both in Combination With Trastuzumab and Capecitabine, for Previously Treated ERBB2 (HER2)-Positive Metastatic Breast Cancer in Patients With Brain Metastases: Updated Exploratory Analysis of the HER2CLIMB Randomized Clinical Trial. JAMA Oncol. 2023 Feb 1;9(2):197-205. doi: 10.1001/jamaoncol.2022.5610. PMID 36454580
- [Derived] Mueller V, Wardley A, Paplomata E, Hamilton E, Zelnak A, Fehrenbacher L, Jakobsen E, Curtit E, Boyle F, Harder Brix E, Brenner A, Crouzet L, Ferrario C, Munoz-Mateu M, Arkenau HT, Iqbal N, Aithal S, Block M, Cold S, Cancel M, Hahn O, Poosarla T, Stringer-Reasor E, Colleoni M, Cameron D, Curigliano G, Siadak M, DeBusk K, Ramos J, Feng W, Gelmon K. Preservation of quality of life in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer treated with tucatinib or placebo when added to trastuzumab and capecitabine (HER2CLIMB trial). Eur J Cancer. 2021 Aug;153:223-233. doi: 10.1016/j.ejca.2021.05.025. Epub 2021 Jun 29. PMID 34214937
- [Derived] Lin NU, Borges V, Anders C, Murthy RK, Paplomata E, Hamilton E, Hurvitz S, Loi S, Okines A, Abramson V, Bedard PL, Oliveira M, Mueller V, Zelnak A, DiGiovanna MP, Bachelot T, Chien AJ, O'Regan R, Wardley A, Conlin A, Cameron D, Carey L, Curigliano G, Gelmon K, Loibl S, Mayor J, McGoldrick S, An X, Winer EP. Intracranial Efficacy and Survival With Tucatinib Plus Trastuzumab and Capecitabine for Previously Treated HER2-Positive Breast Cancer With Brain Metastases in the HER2CLIMB Trial. J Clin Oncol. 2020 Aug 10;38(23):2610-2619. doi: 10.1200/JCO.20.00775. Epub 2020 May 29. PMID 32468955
- [Derived] Murthy RK, Loi S, Okines A, Paplomata E, Hamilton E, Hurvitz SA, Lin NU, Borges V, Abramson V, Anders C, Bedard PL, Oliveira M, Jakobsen E, Bachelot T, Shachar SS, Muller V, Braga S, Duhoux FP, Greil R, Cameron D, Carey LA, Curigliano G, Gelmon K, Hortobagyi G, Krop I, Loibl S, Pegram M, Slamon D, Palanca-Wessels MC, Walker L, Feng W, Winer EP. Tucatinib, Trastuzumab, and Capecitabine for HER2-Positive Metastatic Breast Cancer. N Engl J Med. 2020 Feb 13;382(7):597-609. doi: 10.1056/NEJMoa1914609. Epub 2019 Dec 11. PMID 31825569
- [Derived] Murthy R, Borges VF, Conlin A, Chaves J, Chamberlain M, Gray T, Vo A, Hamilton E. Tucatinib with capecitabine and trastuzumab in advanced HER2-positive metastatic breast cancer with and without brain metastases: a non-randomised, open-label, phase 1b study. Lancet Oncol. 2018 Jul;19(7):880-888. doi: 10.1016/S1470-2045(18)30256-0. Epub 2018 May 24. PMID 29804905

RESULTS

PARTICIPANT FLOW:
Groups:
- Tuc+Cap+Tra: Tucatinib in combination with capecitabine & trastuzumab
- Pbo+Cap+Tra: Placebo in combination with capecitabine & trastuzumab
Period: Overall Study
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Started | 410 | 202
Completed | 0 | 0
Not Completed | 410 | 202
Not completed — Death | 258 | 151
Not completed — Study closure by Sponsor | 119 | 45
Not completed — Withdrawal by Subject | 24 | 5
Not completed — Lost to Follow-up | 7 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Hospital closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Overall Survival (ITT-OS) Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra | Total
Number analyzed (Participants) | 410 | 202 | 612
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 328 | 168 | 496
  >=65 years | 82 | 34 | 116
Age, Continuous [Median (Full Range); unit: years] | 55 [22 to 80] | 54 [25 to 82] | 54 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 407 | 200 | 607
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 14 | 51
  Not Hispanic or Latino | 362 | 184 | 546
  Unknown or Not Reported | 11 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 5 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 41 | 14 | 55
  White | 287 | 157 | 444
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 64 | 26 | 90
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 220 | 111 | 331
  France | 29 | 17 | 46
  United Kingdom | 33 | 12 | 45
  Australia | 27 | 12 | 39
  Canada | 26 | 12 | 38
  Spain | 19 | 7 | 26
  Denmark | 13 | 7 | 20
  Germany | 9 | 8 | 17
  Israel | 13 | 3 | 16
  Belgium | 4 | 6 | 10
  Italy | 6 | 3 | 9
  Austria | 6 | 1 | 7
  Portugal | 3 | 1 | 4
  Czech Republic | 2 | 1 | 3
  Switzerland | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    0: Normal activity | 204 | 94 | 298
    1: Symptoms, but ambulatory | 206 | 108 | 314

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per RECIST 1.1 as Determined by Blinded Independent Central Review (BICR)
Description: Defined as the time from the date of randomization to the date of documented disease progression.
Time Frame: 34.6 months
Population: Intent-to-treat Progression Free Survival (ITT-PFS) Population: Includes the first 480 randomized participants in the ITT analysis population (evaluated by their random treatment assignment).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 320 | 160
months | 7.8 [4.3 to 17.8] | 5.6 [3.0 to 9.7]

2. Secondary Outcome: PFS in Patients With Brain Metastases at Baseline Using RECIST 1.1 as Determined by BICR
Description: Defined as the time from the date of randomization to the date of documented disease progression.
Time Frame: 34.6 months
Population: ITT-PFSBrainMets population: included all randomized participants with brain metastases (evaluated by their random treatment assignment).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 198 | 93
months | 7.6 [4.2 to 11.8] | 5.4 [3.0 to 7.5]

3. Secondary Outcome: Overall Survival (OS) at Time of Primary Analysis
Description: Defined as time from randomization to death from any cause
Time Frame: 35.9 months
Population: ITT-OS Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 410 | 202
months | 21.9 [18.3 to 31.0] | 17.4 [13.6 to 19.9]

4. Secondary Outcome: Confirmed Objective Response Rate (ORR) Per RECIST 1.1 as Determined by BICR
Description: Defined as achieving a best overall response of confirmed complete response (CR) or confirmed partial response (PR).
Time Frame: 34.6 months
Population: ITT - PFS population, subset of participants with measurable disease by BICR at baseline. The ITT-PFS Population includes the first 480 randomized participants in the ITT analysis population (evaluated by their randomized treatment assignment).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 273 | 137
percentage of participants | 40.7 [34.8 to 46.7] | 23.4 [16.6 to 31.3]

5. Secondary Outcome: ORR Per RECIST 1.1 as Determined by Investigator Assessment
Description: Defined as achieving a best overall response of confirmed CR or confirmed PR.
Time Frame: 34.6 months
Population: ITT - PFS population, subset of participants with measurable disease by investigator at baseline. The ITT-PFS Population includes the first 480 randomized participants in the ITT analysis population (evaluated by their randomized treatment assignment).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 280 | 139
percentage of participants | 41.4 [35.6 to 47.4] | 23.0 [16.3 to 30.9]

6. Secondary Outcome: PFS Per RECIST 1.1 as Determined by Investigator Assessment at Time of Primary Analysis
Description: Defined as the time from the date of randomization to the date of documented disease progression
Time Frame: 34.6 months
Population: ITT-PFS Population: Includes the first 480 randomized participants in the ITT analysis population (evaluated by their randomized treatment assignment).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 320 | 160
months | 7.5 [4.1 to 13.1] | 4.3 [2.7 to 8.4]

7. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Determined by BICR
Description: Defined as the time from the first objective response to documented disease progression or death from any cause, whichever occurred first.
Time Frame: 24.6 months
Population: ITT-OS Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 410 | 202
months | 8.3 [4.3 to 12.8] | 6.3 [4.2 to 9.0]

8. Secondary Outcome: DOR Per RECIST 1.1 as Determined by Investigator Assessment
Description: as for outcome 7
Time Frame: 33.2 months
Population: ITT-OS Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 410 | 202
months | 7.0 [4.3 to 12.9] | 6.9 [4.1 to 9.6]

9. Secondary Outcome: Clinical Benefit Rate (CBR) as Determined by BICR Per RECIST 1.1
Description: Clinical benefit was defined as achieving stable disease (SD) or non-complete response (CR)/non-progressive disease (PD) for at least 6 months or a best overall response of confirmed CR or confirmed partial response (PR).
Time Frame: 34.6 months
Population: ITT-OS Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 410 | 202
percentage of participants | 59.8 [54.8 to 64.5] | 38.1 [31.4 to 45.2]

10. Secondary Outcome: CBR Per RECIST 1.1 as Determined by Investigator Assessment
Description: Clinical benefit was defined as achieving stable disease (SD) or non-CR/non-PD for at least 6 months or a best overall response of confirmed CR or confirmed PR.
Time Frame: 34.6 months
Population: ITT-OS Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 410 | 202
percentage of participants | 58.0 [53.1 to 62.9] | 37.6 [30.9 to 44.7]

11. Secondary Outcome: Incidence of Adverse Events (AEs) at Time of Primary Analysis
Description: As determined by assessment of AEs, clinical laboratory tests, and vital signs measurements. AEs were classified by system organ class (SOC) and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA) Version 22.0 or higher; AE severities were classified using Version 4.03 of the (Common Terminology Criteria for Adverse Events) CTCAE criteria.
Time Frame: 36.1 months
Population: Safety Analysis Population: Includes all randomized participants who received at least one dose of study treatment (tucatinib/placebo, trastuzumab, or capecitabine), with participants allocated to the treatment group associated with the regimen actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 404 | 197
Participants
  Any treatment-emergent AE (TEAE) | 401 | 191
  Any Grade 3 or higher TEAE | 223 | 96
  Any treatment-emergent serious AE | 104 | 53
  TEAE leading to death | 8 | 6

12. Secondary Outcome: Frequency of Dose Modifications
Time Frame: 35.1 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 404 | 197
Participants
  TEAEs resulting in tuc/pbo dose modification | 220 | 81
  TEAEs resulting in tucatinib/placebo dose hold | 216 | 80
  TEAEs resulting in tuc/pbo dose reduction | 84 | 21
  TEAEs resulting capecitabine dose modification | 313 | 122
  TEAEs resulting in capecitabine dose hold | 276 | 113
  TEAEs resulting in capecitabine dose reduction | 243 | 77
  TEAEs resulting trastuzumab dose modification | 104 | 38
  TEAEs resulting in trastuzumab dose hold | 104 | 38

13. Secondary Outcome: Incidence of Health Resources Utilization
Description: Cumulative incidence of health resource utilization, including length of stay, hospitalizations, and ER visits using the EQ-5D-5L questionnaire.
Time Frame: 36.1 months
Population: as for outcome 11
Measure: Number; unit: hospitalizations
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 404 | 197
hospitalizations
  Total number of hospitalizations | 143 | 75
  Hospitalization for AE | 124 | 64
  Planned hospitalization (other than AE) | 10 | 6
  Ambulatory Surgery | 3 | 0
  Other | 6 | 5

14. Secondary Outcome: Pharmacokinetic Measure: Ctrough of Tucatinib
Description: Individual plasma tucatinib concentrations at each sampling time
Time Frame: 3.5 months
Population: Pharmacokinetics (PK) Analysis Set: Includes all randomized participants who received at least one dose of tucatinib and who had at least one evaluable PK assessment. Participants were evaluated by the treatment actually received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tuc+Cap+Tra
Number analyzed (Participants) | 373
ng/mL
  Cycle 2, Day 1 (Pre-dose) | 246.1 (260.9)
  Cycle 3, Day 1 (Pre-dose) | 227.6 (210.8)
  Cycle 3, Day 1 (Post-dose) | 507.1 (357.1)
  Cycle 4, Day 1 (Pre-dose) | 253.2 (236.1)
  Cycle 5, Day 1 (Pre-dose) | 257.6 (286.9)
  Cycle 6, Day 1 (Pre-dose) | 247.8 (225.1)

15. Secondary Outcome: Pharmacokinetic Measure: ONT-993
Description: Individual plasma primary metabolite concentrations at each sampling time
Time Frame: 3.5 months
Population: PK Analysis Set: Includes all randomized participants who received at least one dose of tucatinib and who had at least one evaluable PK assessment. Participants were evaluated by the treatment actually received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tuc+Cap+Tra
Number analyzed (Participants) | 373
ng/mL
  Cycle 2, Day 1 (Pre-dose) | 25.5 (24.4)
  Cycle 3, Day 1 (Pre-dose) | 22.6 (20.6)
  Cycle 3, Day 1 (Post-dose) | 47.7 (47.2)
  Cycle 4, Day 1 (Pre-dose) | 25.2 (24.3)
  Cycle 5, Day 1 (Pre-dose) | 24.5 (30.6)
  Cycle 6, Day 1 (Pre-dose) | 20.9 (18.0)

16. Secondary Outcome: Overall Survival (OS) at Time of Final Analysis
Description: Defined as time from randomization to death from any cause
Time Frame: Up to 60.1 months
Population: ITT-OS Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 410 | 202
months | 24.7 [21.6 to 28.9] | 19.2 [16.4 to 21.4]

17. Secondary Outcome: PFS Per RECIST 1.1 as Determined by Investigator Assessment at Time of Final Analysis
Description: Defined as the time from the date of randomization to the date of documented disease progression
Time Frame: Up to 58.0 months
Population: ITT-OS Population: Includes all randomized participants evaluated by their randomized treatment assignment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 410 | 202
months | 7.6 [4.1 to 13.8] | 4.9 [2.7 to 9.0]

18. Secondary Outcome: Incidence of Adverse Events (AEs) at Time of Final Analysis
Description: as for outcome 11
Time Frame: Up to 60.1 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 404 | 197
Participants
  Any treatment-emergent AE (TEAE) | 401 | 191
  Any Grade 3 or higher TEAE | 248 | 101
  Any treatment-emergent serious AE | 123 | 58
  TEAE leading to death | 8 | 6

19. Secondary Outcome: Frequency of Dose Modifications at Time of Final Analysis
Time Frame: Up to 60.1 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
Number analyzed (Participants) | 404 | 197
Participants
  TEAEs resulting in tuc/pbo dose modification | 237 | 85
  TEAEs resulting in tucatinib/placebo dose hold | 232 | 84
  TEAEs resulting in tuc/pbo dose reduction | 92 | 21
  TEAEs resulting capecitabine dose modification | 322 | 125
  TEAEs resulting in capecitabine dose hold | 288 | 117
  TEAEs resulting in capecitabine dose reduction | 251 | 79
  TEAEs resulting trastuzumab dose modification | 117 | 41
  TEAEs resulting in trastuzumab dose hold | 117 | 41

ADVERSE EVENTS:
Time Frame: Non-serious Adverse Events, Serious Adverse Events, and All-Cause Mortality were followed for up to 60.1 months
Arm/Group | Tuc+Cap+Tra | Pbo+Cap+Tra
All-Cause Mortality (participants affected / at risk) | 262/410 | 152/202
Serious Adverse Events (participants affected / at risk) | 124/404 | 62/197
Other Adverse Events (participants affected / at risk) | 399/404 | 188/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tuc+Cap+Tra (N=404) | Pbo+Cap+Tra (N=197)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 7 (8)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (10) | 4 (4)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (12) | 5 (5)
Fatigue (General disorders) | 3 (3) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Sudden death (General disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (9) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Septic shock (Infections and infestations) | 1 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2)
Ejection fraction decreased (Investigations) | 6 (6) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 2 (2)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (2) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 11 (11) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 6 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tuc+Cap+Tra (N=404) | Pbo+Cap+Tra (N=197)
Anaemia (Blood and lymphatic system disorders) | 89 (146) | 24 (32)
Neutropenia (Blood and lymphatic system disorders) | 37 (87) | 17 (40)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (41) | 11 (15)
Dry eye (Eye disorders) | 23 (25) | 10 (10)
Abdominal distension (Gastrointestinal disorders) | 27 (30) | 10 (13)
Abdominal pain (Gastrointestinal disorders) | 66 (98) | 32 (40)
Abdominal pain upper (Gastrointestinal disorders) | 36 (43) | 17 (20)
Constipation (Gastrointestinal disorders) | 69 (90) | 40 (46)
Diarrhoea (Gastrointestinal disorders) | 330 (812) | 106 (181)
Dry mouth (Gastrointestinal disorders) | 22 (22) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 46 (53) | 19 (22)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 25 (27) | 7 (7)
Nausea (Gastrointestinal disorders) | 243 (382) | 87 (120)
Stomatitis (Gastrointestinal disorders) | 105 (146) | 28 (35)
Vomiting (Gastrointestinal disorders) | 155 (276) | 49 (80)
Asthenia (General disorders) | 34 (46) | 15 (19)
Fatigue (General disorders) | 193 (265) | 87 (108)
Influenza like illness (General disorders) | 24 (31) | 6 (6)
Oedema peripheral (General disorders) | 46 (52) | 19 (25)
Pyrexia (General disorders) | 25 (35) | 8 (10)
Hyperbilirubinaemia (Hepatobiliary disorders) | 29 (69) | 8 (17)
Influenza (Infections and infestations) | 10 (10) | 10 (10)
Nasopharyngitis (Infections and infestations) | 21 (28) | 14 (15)
Paronychia (Infections and infestations) | 23 (30) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 45 (70) | 15 (18)
Urinary tract infection (Infections and infestations) | 45 (76) | 16 (24)
Fall (Injury, poisoning and procedural complications) | 28 (41) | 9 (10)
Alanine aminotransferase increased (Investigations) | 87 (115) | 13 (15)
Aspartate aminotransferase increased (Investigations) | 92 (137) | 23 (32)
Blood alkaline phosphatase increased (Investigations) | 29 (47) | 6 (8)
Blood bilirubin increased (Investigations) | 81 (154) | 21 (31)
Blood creatinine increased (Investigations) | 65 (108) | 3 (3)
Neutrophil count decreased (Investigations) | 21 (48) | 6 (7)
Platelet count decreased (Investigations) | 22 (29) | 5 (6)
Weight decreased (Investigations) | 62 (66) | 12 (13)
White blood cell count decreased (Investigations) | 21 (57) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 108 (130) | 41 (51)
Dehydration (Metabolism and nutrition disorders) | 31 (40) | 10 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 26 (40) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 71 (105) | 24 (32)
Hypomagnesaemia (Metabolism and nutrition disorders) | 37 (61) | 10 (10)
Hypophosphataemia (Metabolism and nutrition disorders) | 29 (50) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 (120) | 17 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 58 (73) | 25 (27)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 46 (63) | 6 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 22 (25) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 34 (43) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 (66) | 18 (22)
Dizziness (Nervous system disorders) | 54 (68) | 27 (30)
Dysgeusia (Nervous system disorders) | 33 (33) | 6 (6)
Headache (Nervous system disorders) | 98 (150) | 38 (53)
Paraesthesia (Nervous system disorders) | 26 (32) | 10 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 53 (65) | 13 (17)
Insomnia (Psychiatric disorders) | 40 (45) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 67 (85) | 24 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 53 (60) | 23 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 52 (63) | 10 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 31 (37) | 9 (14)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 28 (32) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 25 (26) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 43 (53) | 18 (20)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 265 (433) | 105 (158)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (48) | 15 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 (43) | 10 (13)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 34 (45) | 11 (11)
Hypertension (Vascular disorders) | 19 (30) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT02614794/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT02614794/SAP_003.pdf